CLINICAL TRIAL: NCT04403048
Title: Rationale and Design of a Prospective, Open Label, Randomized, Multicentric Clinical Trial: Drug Coated Balloon for Side Branch Treatment vs. Conventional Approach in True Bifurcation Coronary Disease: PRO-DAVID
Brief Title: Drug Coated Balloon for Side Branch Treatment vs. Conventional Approach in True Bifurcation Coronary Disease: PRO-DAVID
Acronym: PRO-DAVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Deiti Prvulovic, Principal Investigator, MD, PhD, Clinical Hospital Center Rijeka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-DAVID
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Stable Angina; Ischemic Heart Disease; Coronary Artery Disease; Unstable Angina; NSTEMI - Non-ST Segment Elevation MI
Keywords: Drug Coated Ballon; Bifurcation coronary disease; SYNTAX score; Medina classification; Coronary angiography
MeSH Terms: conditions — Angina, Stable; Myocardial Ischemia; Coronary Artery Disease; Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in which standard provisional approach is preformed (Active Comparator): Detailed technique is described in the Detailed study description paragraph
  Interventions: Procedure: Standard provisional approach PCI procedure
- Patients in which provisional DCB approach is preformed (Experimental): Detailed technique is described in the Detailed study description paragraph
  Interventions: Procedure: Provisional DCB approach PCI procedure

INTERVENTIONS:
Procedure: Provisional DCB approach PCI procedure — Intervention is explained in detail in group description
  Arms: Patients in which provisional DCB approach is preformed
Procedure: Standard provisional approach PCI procedure — Intervention is explained in detail in group description
  Other Names: any 2-stent technique for bail-out patients
  Arms: Patients in which standard provisional approach is preformed

SUMMARY:
Bifurcation lesions (BL) on coronary arteries account for 15-20 % of all performed percutaneous coronary interventions (PCI). Preferred approach for treatment of most bifurcation lesions is the stepwise provisional stent strategy with main branch-only stenting followed by provisional balloon angioplasty with or without stenting of the side branch (SB). Stenting of the side branch is indicated when the angiographic result in SB is clearly suboptimal and when flow remains reduced. Upfront use of two stent techniques may be indicated in very complex lesions with large calcified side branches ( most likely to supply at least 10% of fractional myocardial mass), with a long ostial side branch lesion (>5mm) or anticipated difficulty in accessing an important side branch after main branch stenting, and true distal LM bifurcations.

From a technical point of view, we propose a "Provisional DCB approach" that differs from the standard provisional approach with obligatory SB predilation and good lesion preparation. In case of an adequate result of predilation, the procedure on the SB ends with the DCB deployment. This is followed by main branch stenting with DES, finished with POT. Final 'kissing' balloon dilation is generally not recommended because there is no advantage from final kissing with the one-stent technique. With this approach, there is no need for re-wiring, re-ballooning, side branching and wire jailing and final kissing. This technique is close to a contemporary approach to bifurcation lesions based on the fundamental philosophy of the European Bifurcation Club (EBC): keep it simple, systematic, and safe, with a limited number of stents that should be well apposed and expanded with limited overlap, with respect of the original bifurcation anatomy.

DETAILED DESCRIPTION:
Bifurcation lesions (BL) on coronary arteries account for 15-20 % of all performed percutaneous coronary interventions (PCI). Preferred approach for treatment of most bifurcation lesions is the stepwise provisional stent strategy with main branch-only stenting followed by provisional balloon angioplasty with or without stenting of the side branch (SB). Stenting of the side branch is indicated when the angiographic result in SB is clearly suboptimal and when flow remains reduced. Upfront use of two stent techniques may be indicated in very complex lesions with large calcified side branches ( most likely to supply at least 10% of fractional myocardial mass), with a long ostial side branch lesion (>5mm) or anticipated difficulty in accessing an important side branch after main branch stenting, and true distal LM bifurcations.

For non-left main bifurcation lesions consensus is that there is no systematic advantage to a more complex dual-stent implantation technique. For true left main lesions EAPCI/EACTS revascularization guidelines gave a IIb recommendation for double-kissing crush two-stent strategy compared to the provisional approach, based on the results of DKCRUSH-V Trial. EBC perspectives, even for the stenting on left main coronary true bifurcation lesions, is that they are best treated with a planned single-stent strategy rather than a planned dual-stent strategy. When a two-stent strategy is used, this will become apparent during a provisional stepwise approach, and finalizing the procedure using a culotte technique or occasionally TAP is recommended.

PCI strategies for complex coronary bifurcation lesions should be individualized, taking into account the anatomical differentiation of coronary bifurcation lesion differences, disease burden and complexity, but also the technical skills and experience of the operator. In daily clinical practice where less experienced operators with limited number of true bifurcations annually are faced with the challenge of treating complex bifurcation lesions, it is imperative to find a standardized and universal approach which would be simple, quick and safe, with a high percentage of procedural success, with a small number of complications, good long term results, with small expenditure of material and contrast volumes, and shorter procedure and fluoroscopy times.

Drug-coated balloon (DCB) technology allows to bring high concentration of an antiproliferative drug with immediate and rapid local delivery even with short contact times between the balloon surface and the vessel wall, sufficient for effective drug delivery without a durable polymer and further permanent metal prosthesis. The application of DCB in SB is an attractive and intriguing solution in treating complex BL. Rationality of such an approach lies in the many theoretical advantages of DCB. The application of DCB in SB respects the original anatomy of bifurcation, which is especially important in the carina area, and allows for the homogeneous application of a high dose of antiproliferative drug on the entire blood vessel surface and avoids the risk of incomplete coverage of the bifurcation area. In the case of a successful DCB application in the SB, unnecessary use of the stent is avoided, obviating long-term problems such as stent malposition and fracturing, scaffolding of the SB ostium, overlapping and crushing of multiple metal layers and polymers with uncontrolled drug release, and therefore re-stenosis and thrombosis and reactions to a foreign body. Even for the simplest provisional technique, the application of DCB has a theoretical advantage over the application of a regular balloon, with the expected positive remodelling of the vessel and plaque stabilization, and better late angiographic results, as well as neoatherosclerosis.

From a technical point of view, we propose a "Provisional DCB approach" that differs from the standard provisional approach with obligatory SB predilation and good lesion preparation. In case of an adequate result of predilation, the procedure on the SB ends with the DCB deployment. This is followed by main branch stenting with DES, finished with POT. Final 'kissing' balloon dilation is generally not recommended because there is no advantage from final kissing with the one-stent technique. With this approach, there is no need for re-wiring, re-ballooning, side branching and wire jailing and final kissing. This technique is close to a contemporary approach to bifurcation lesions based on the fundamental philosophy of the European Bifurcation Club (EBC): keep it simple, systematic, and safe, with a limited number of stents that should be well apposed and expanded with limited overlap, with respect of the original bifurcation anatomy.

The study hypothesis is that in patients with true complex bifurcation lesions (Medina 1,1,1; 1,0,1; 0,1,1) with significant SB, intervention using DCB first in SB and DES in the main vessel will not be inferior then planned single-stent strategy treating with superiority in the simplicity of procedure.

The registry will include patients requiring percutaneous coronary interventions with true bifurcation lesions (Medina 1,1,1; 1,0,1; 0,1,1) of unprotected left main coronary bifurcation disease, and non left main bifurcational lesion with affected important side branches most likely to supply at least 10% of fractional myocardial mass. The SYNTAX score for the lesions that are to be treated should be <32.

Patients who fulfill inclusion and exclusion criteria and consent to the study will be randomized according to a standard random number generation method. Patient randomisation will be stratified by participating centre.

A diagnostic coronary angiography will be performed on all patients who have the clinical criteria for inclusion into the trial. All of the procedures will be carried out by classical radial or femoral approach depending on the operator choice, and the intervention will be carried out ad hoc or electively, at the operator discretion. Before the PCI procedure the patients will receive 300 mg of acetylsalicylic acid (100 mg if they were saturated earlier) 600 mg clopidogrel (75 mg if they were saturated earlier), or 2 x 90 mg ticagrelor and unfractionated heparin 70 - 100 UI/kg of body weight. The administration of intergrilin is upon operator decision. After intracoronary application of 100-200 µg of nitroglycerin a diagnostic angiogram will be carried out to record several views from various angles to obtain an optimal angiographic view that allows the visualization of branch division as well as the measurement of angles and assessment of the degree of ostial SB stenosis , "the working view". Planned single- and dual-stent techniques will be performed according to the recommendation of the EBC consensus.

The patients will be randomized in one of two groups including standard provisional approach or provisional DBC approach.

Standard provisional approach technique:

Coronary guidewires should be passed to the both main branch ( MB ) and side branch ( SB ) vessels. MB preparation should be considered routine practice in stable patients, but initial SB predilatation is only recommended when access is difficult, in cases of severe diffuse and/or calcified SB lesion or compromised SB flow after wiring. Stenting of the main vessel should be undertaken with a wire jailed in the side vessel to preserve side vessel flow and access. Second-generation DES should be used and stent diameter should be chosen according to the size of the MB beyond the bifurcation, and according to the expansion ability of the stent in proximal MB with proximal optimisation technique ( POT ). Following stenting of the MB, POT should be performed routinely with a short appropriately sized non-compliant balloon. Following POT, rewiring of the SB should aim to recross a distal stent cell. KBI should be performed using two NC balloons, sized according to the actual reference size of the vessels or 0.5 mm below, with individual high-pressure inflation followed by a final lower-pressure kiss dilatation. The procedure should be finalised by POT after kissing to correct the proximal MB stent distortion. SB should not be treated further unless there is one of the following: TIMI flow <3 in the SB, severe ostial pinching of SB(>90%), threatened SB closure, SB vessel dissection >type A, or FFR > 0,80. Bail-out SB stenting after MB stenting is performed with T-stenting, T and protrusion ( TAP ) or culotte. Implantation technique is selected according to angulations, reference size differences and operator capabilities. If SB stenting is necessary, it should be followed by KBI, and the procedure should be finalised with a second POT

Provisional DCB approach:

Wiring of MB and SB and MB preparation is the same as in standard provisional approach. Initial SB predilatation is obligatory. Predilatation of SB is done with semicompliant or noncompliant balloon, with balloon to vessel ratio of 0.8-1:1 at nominal inflation pressures. Liberal use of scoring or cutting balloons sized 0.5 mm smaller than the vessel size and inflated to high pressure is also recommended. Angio check is repeated after 10 minutes and intracoronary nitroglycerin application to rule out acute recoil. DCB is inflated in SB only after successful predilatation defined as residual stenosis ≤ 30% and no C,D,E,F dissection. Manipulation of the DCB should be done in the way to avoid drug loss during transit : no manipulation during flushing, lesion site should be reached rapidly, care should be taken when crossing the Y-connector and navigating through the proximal coronary artery up to the lesion. Inflation time when applying a DCB is 60 s, using DCB to vessel ratio of 0.8-1:1 at low inflation pressures that should not exceed nominal pressure, to reduce the risk of dissection. DCB inflation in SB is followed by a DES deployment in the main branch. POT is mandatory, and a final kissing balloon or POT/side/POT is not done.

Bail out stenting of SB could be done at two points of the procedure. First decision on the need for bail out SB stenting is after predilatation of SB and angio check. Bail out stenting is indicated in case of unsuccessful SB predilatation ( dissection C,D,E,F, or residual stenosis >30% ) or in case of decreased flow-TIMI <3, acute recoil, ischemia or FFR > 0,80. Bail-out SB stenting can be performed with any two stent technique. Implantation technique is selected according to angulations, reference size differences and operator capabilities, followed by KBI, and the procedure should be finalised with a second POT. After deployment of DCB and POT, there is second decision to perform bail out SB stenting. Here it is indicated in SB pinching ≥ 90% stenosis or FFR > 0,80 , dissection >type A, threatened SB closure, decreased flow - TIMI <3 or ischemia. Bail-out SB stenting after MB stenting is performed with T-stenting, T and protrusion ( TAP ) or culotte. Implantation technique is selected according to angulations, reference size differences and operator capabilities. If SB stenting is necessary, it should be followed by KBI, and the procedure should be finalised with a second POT.

Patients will be followed up by telephone or in person 1, 6, 12 and 36 months, and optional angiographical control after 9 months.

Significant symptoms will trigger further investigation as required.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the inclusion criteria:

Clinical:

1. stable angina Canadian Cardiovascular Society (CCS) 2 to 4, unstable angina, NSTEMI
2. clinical and anatomic eligibility for PCI as agreed to by the local Heart Team
3. in stable angina: a. ischaemic symptoms, or b. proof of ischemia on nonvasive testing, or c. positive FFR or iFR or d. ( for LMS ) IVUS minimal lumen area <6 mm²
4. patients with mental and logistical conditions for further monitoring
5. patients need to accept clinical monitoring during 3 years and sign a written consent form
6. patients need to be older than 18 years

Angiographical:

1. de novo bifurcational lesion with affected side branch (Medina 1,1,1; 1,0,1; 0,1,1)
2. side branch diameter ≥ 2,5 mm
3. LM SB-DS ≥70% and SB lesion length > 5 mm
4. non LM: SB-DS ≥ 90% and SB lesion length > 5 mm
5. side branch length ≥ 73mm
6. for patients with LAD/diagonal BL - Scoring system for diagonal branches (Modified SNuHscore) ≥ 2

Exclusion Criteria:

Clinical:

1. STEMI <72 hours preceding
2. Chronic total occlusion of either vessel
3. SYNTAX score for planned lesions to be treated >32
4. cerebrovascular accident within 6 months, surgical procedure within one week
5. pregnant/nursing women
6. ejection fraction LV< 30%, congestive heart failure, cardiogenic shock or sever valvular disease
7. unfavourable long-term prognosis - patient life expectancy less than 12 months
8. creatinine > 2,0 mg/dl ( 177 mmol/L)
9. hypersensibility, allergies or contraindication to: aspirin, heparin, clopidogrel, prasugel, steel, sirolimus, everolimus, zotarolimus, biolimus or contrast agents
10. treatment of hyperthyroidism, administration of immunosuppressives or anticoagulant therapy, addiction to alcohol or drugs
11. patients included in other clinical trials

Angiographical:

1. thrombotic lesions
2. severe calcification
3. patients who have had a stent implanted previously ≤ 15 mm from the current lesions which is included in the study
4. lesions on the aorto-coronary venous or arterial grafts or on chronic total occlusions
5. In-stent restenosis or restenosis in a segment closer than 4 mm from the target lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop major adverse cardiac events | 12 months after the procedure
  Defined as cardiac death, myocardial infarction unrelated to the procedure which demanded hospitalization, revascularization of the target lesion

SECONDARY OUTCOMES:
Number of patients who develop an individual component of the primary endpoint | 12 months and 36 months after the procedure
  cardiac death, myocardial infarction unrelated to the procedure which demanded hospitalization, revascularization of the target lesion
Rate of angiographic success | immediately after the procedure
  residual stenosis - main blood vessel ≤10%, side branch vessel: ≤30%, visual assessment of quantitative angiography, TIMI 3 flow in both treated blood vessels, no flow-limiting dissection, distal embolization or thrombus seen on angiography
Rate of procedural success | immediately after the procedure
  angiographic success without intrahospital MACE which include death, infarction with ST elevation or emergency bypass surgery
Rate of possible, probable or definitive stent thrombosis | 12 months after the procedure
  ARC definition
Rate of in segment late lumen loss in any of the treated branches | 9 months after the procedure
  standard definition
Rate of "bailout" stenting and inadequate predilatation | immediately after the procedure
  standard definition
Fluoroscopy time | immediately after the procedure
  standard definition
Fluoroscopy dose | immediately after the procedure
  standard definition
Contrast volume | immediately after the procedure
  standard definition
Assessing a composite of the number of guidewires, balloons and stents opened or used | immediately after the procedure
  standard definition
Rate lumen gain difference of 20% | 6-9 months after the procedure
  measured by IVUS or OCT

CONTACTS AND LOCATIONS:
Overall Officials: Deiti Prvulovic, MD, PhD, Principal Investigator — Clinical Hospital Center Rijeka

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Latib A, Colombo A. Bifurcation disease: what do we know, what should we do? JACC Cardiovasc Interv. 2008 Jun;1(3):218-26. doi: 10.1016/j.jcin.2007.12.008. PMID 19463303
- [Background] Meier B, Gruentzig AR, King SB 3rd, Douglas JS Jr, Hollman J, Ischinger T, Aueron F, Galan K. Risk of side branch occlusion during coronary angioplasty. Am J Cardiol. 1984 Jan 1;53(1):10-4. doi: 10.1016/0002-9149(84)90675-1. PMID 6229173
- [Background] Myler RK, Shaw RE, Stertzer SH, Hecht HS, Ryan C, Rosenblum J, Cumberland DC, Murphy MC, Hansell HN, Hidalgo B. Lesion morphology and coronary angioplasty: current experience and analysis. J Am Coll Cardiol. 1992 Jun;19(7):1641-52. doi: 10.1016/0735-1097(92)90631-v. PMID 1593061
- [Background] Lefevre T, Louvard Y, Morice MC, Dumas P, Loubeyre C, Benslimane A, Premchand RK, Guillard N, Piechaud JF. Stenting of bifurcation lesions: classification, treatments, and results. Catheter Cardiovasc Interv. 2000 Mar;49(3):274-83. doi: 10.1002/(sici)1522-726x(200003)49:33.0.co;2-n. PMID 10700058
- [Background] Banning AP, Lassen JF, Burzotta F, Lefevre T, Darremont O, Hildick-Smith D, Louvard Y, Stankovic G. Percutaneous coronary intervention for obstructive bifurcation lesions: the 14th consensus document from the European Bifurcation Club. EuroIntervention. 2019 May 20;15(1):90-98. doi: 10.4244/EIJ-D-19-00144. PMID 31105066
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Chen SL, Zhang JJ, Han Y, Kan J, Chen L, Qiu C, Jiang T, Tao L, Zeng H, Li L, Xia Y, Gao C, Santoso T, Paiboon C, Wang Y, Kwan TW, Ye F, Tian N, Liu Z, Lin S, Lu C, Wen S, Hong L, Zhang Q, Sheiban I, Xu Y, Wang L, Rab TS, Li Z, Cheng G, Cui L, Leon MB, Stone GW. Double Kissing Crush Versus Provisional Stenting for Left Main Distal Bifurcation Lesions: DKCRUSH-V Randomized Trial. J Am Coll Cardiol. 2017 Nov 28;70(21):2605-2617. doi: 10.1016/j.jacc.2017.09.1066. Epub 2017 Oct 30. PMID 29096915
- [Background] Chieffo A, Hildick-Smith D. The European Bifurcation Club Left Main Study (EBC MAIN): rationale and design of an international, multicentre, randomised comparison of two stent strategies for the treatment of left main coronary bifurcation disease. EuroIntervention. 2016 May 17;12(1):47-52. doi: 10.4244/EIJV12I1A8. PMID 27173861
- [Background] Ann SH, Balbir Singh G, Lim KH, Koo BK, Shin ES. Anatomical and Physiological Changes after Paclitaxel-Coated Balloon for Atherosclerotic De Novo Coronary Lesions: Serial IVUS-VH and FFR Study. PLoS One. 2016 Jan 29;11(1):e0147057. doi: 10.1371/journal.pone.0147057. eCollection 2016. PMID 26824602
- [Background] Her AY, Ann SH, Singh GB, Kim YH, Yoo SY, Garg S, Koo BK, Shin ES. Comparison of Paclitaxel-Coated Balloon Treatment and Plain Old Balloon Angioplasty for De Novo Coronary Lesions. Yonsei Med J. 2016 Mar;57(2):337-41. doi: 10.3349/ymj.2016.57.2.337. PMID 26847284
- [Background] Niemela M, Kervinen K, Erglis A, Holm NR, Maeng M, Christiansen EH, Kumsars I, Jegere S, Dombrovskis A, Gunnes P, Stavnes S, Steigen TK, Trovik T, Eskola M, Vikman S, Romppanen H, Makikallio T, Hansen KN, Thayssen P, Aberge L, Jensen LO, Hervold A, Airaksinen J, Pietila M, Frobert O, Kellerth T, Ravkilde J, Aaroe J, Jensen JS, Helqvist S, Sjogren I, James S, Miettinen H, Lassen JF, Thuesen L; Nordic-Baltic PCI Study Group. Randomized comparison of final kissing balloon dilatation versus no final kissing balloon dilatation in patients with coronary bifurcation lesions treated with main vessel stenting: the Nordic-Baltic Bifurcation Study III. Circulation. 2011 Jan 4;123(1):79-86. doi: 10.1161/CIRCULATIONAHA.110.966879. Epub 2010 Dec 20. PMID 21173348
- [Background] Gwon HC, Hahn JY, Koo BK, Song YB, Choi SH, Choi JH, Lee SH, Jeong MH, Kim HS, Seong IW, Yang JY, Rha SW, Jang Y, Yoon JH, Tahk SJ, Seung KB, Park SJ. Final kissing ballooning and long-term clinical outcomes in coronary bifurcation lesions treated with 1-stent technique: results from the COBIS registry. Heart. 2012 Feb;98(3):225-31. doi: 10.1136/heartjnl-2011-300322. Epub 2011 Sep 20. PMID 21933939